CLINICAL TRIAL: NCT02926456
Title: Italian Observational, Multicenter Study in HIV1 -Positive, Virosuppressed Patients Currently in Treatment With Ritonavir-boosted Protease Inhibitors (PI/r) Starting Cobicistat-boosted Darunavir (DRV/c - Rezolsta®): the STart Of REzolsta (ST.O.RE.) Study
Brief Title: Study in HIV1-Positive, Virosuppressed Patients Currently inTreatment With Ritonavir-Boosted Protease Inhibitors (PI/r) Starting Cobicistat-Boosted Darunavir (DRV/c - Rezolsta)
Acronym: STORE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108148; TMC114FD1HTX4003 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2016-09-21; First posted 2016-10-06 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: HIV-1-infected patients being in stable ritonavir-boosted Antiretroviral (ARV) treatment with Protease Inhibitors (PIs) (either darunavir 800 milligram [mg] each day -based or not) since at least twelve months and virologically suppressed (HIV-RNA less than [<]50 copies/milliliters) since at least six months.

SUMMARY:
The purpose of this study is to describe the effectiveness of darunavir/cobicistat (DRV/c)-based regimens, measured as maintenance of virological suppression 48 weeks after baseline, defined as the day when the treatment with DRV/c-based regimen is started, through collection of daily practice data in the Italian setting.

ELIGIBILITY:
Inclusion Criteria:

* Adult greater than or equal to (>=18 years), male and female patients
* Documented Human Immunodeficiency Virus-1 (HIV-1) infection
* Eligible to darunavir/cobicistat (DRV/c) treatment according to Summary of Product Characteristics
* Patients who are able to understand the nature of the study and to provide their consent voluntarily having signed an Informed Consent Form (ICF) allowing data collection and source data verification in accordance with local requirements
* Patients in stable (>= 12 months) treatment with an Antiretroviral (ARV) therapy PI/ritonavir (PI/r)-based, being prescribed Rezolsta (DRV/c) by treating physician
* Patients virosuppressed (HIV-RNA less than [<] 50 copies/milliliters) since at least 6 months, within their HIV treatment at the moment of enrollment; single values of HIV-RNA more than [>] 50 copies/ml not confirmed (blips) will be considered acceptable; last value collected being < 50 copies/ml

Exclusion Criteria:

* Patient currently enrolled in an interventional study
* Patient currently enrolled in an observational study sponsored or supported by Janssen
* Estimated Glomerular Filtration Rate (eGFR) < 70 milliliters per minute (ml/min) if any co-administered agent (example emtricitabine, lamivudine, tenofovir disoproxil fumarate, or adefovir dipivoxil) requires dose adjustment based on creatinine clearance
* Pregnancy or breast feeding at enrollment
* Allergy or intolerance to sulphonamides
* Switch from darunavir/ritonavir (DRV/r) 600/100 bis in die (bid)
* Patient currently in mono PI/r therapy
* Patients to be treated within one year with Direct Acting Antivirals (DAAs) for Hepatitis C Virus (HCV) infection
* Chemotherapy scheduled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult out-patients with a confirmed diagnosis of Human Immunodeficiency Virus-1 (HIV-1), belonging to Italian Infectious Disease Hospital departments of Italian specialty hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients With Human Immunodeficiency Virus - RiboNucleic Acid (HIV-RNA) Less Than (<)50 Copies/Milliliters (copies/mL) Measured at Week 48 | At Visit 4 (Week 48)
  The percentage of patients with plasma HIV-RNA<50 copies/mL will be analyzed by FDA snapshot analysis (FDA Snapshot Approach is based on the last observed viral load data within the Week 48 window: virologic response is defined as HIV-1 RNA <50 copies/mL (observed case); If there are no data in the defined time window, the proportion of missing data and relative reason will be provided") and Time to loss of virologic response (TLOVR) method algorithm requires sustained HIV-1 RNA < 50 copies/mL; confirmed HIV-1 RNA more than or equal to (>=) 50 copies/mL is considered as non-response (rebound); patients considered non-responder after permanent discontinuation).

SECONDARY OUTCOMES:
Change From Baseline in HIV-Symptoms Distress Module (HIV-SDM) Score | Baseline, Up to Visit 4 (Week 48)
  HIV-SDM is a questionnaire consisting of 20 questions related to all the symptoms which the patient might have had during the past four weeks. For each question patient has to select appropriate answer related to the symptoms: "0 = I do not have this symptom; 1 = I have this symptom and it doesn't bother me; 2 = it bothers me a little; 3 = it bothers me; 4 = it bothers me a lot".
Change From Baseline in HIV-Treatment Satisfaction Questionnaire (HIV-TSQ) Score | Baseline, Up to Visit 4 (Week 48)
  The HIV Treatment Satisfaction Questionnaire (HIV-TSQ) is a 10-item instrument that is supported by evidence of good internal consistency reliability. The total score ranges from 0 to 60, with higher scores indicating greater treatment satisfaction. Score change ranges from -30 to +30, with scores<0 and >0 indicating a decrease and increase in treatment satisfaction, respectively.
Percentage of Patients with HIV-RNA <50 copies/mL Measured at Week 24 | At Visit 3 (Week 24)
Change From Baseline in CD4 Cell Count | Baseline, Up to Visit 4 (Week 48)
  CD4 cell count will be assessed as immunological parameter.
Change From Baseline in CD4/CD8 Ratio | Baseline, Up to Visit 4 (Week 48)
  CD4/CD8 ratio will be assessed as immunological parameter.
Change From Baseline in CD4 Percentage | Baseline, Up to Visit 4 (Week 48)
  CD4 percentage will be assessed as immunological parameter.
Change From Baseline in Creatinine Levels | Baseline, Up to Visit 4 (Week 48)
  The change from baseline in serum creatinine up to 48 weeks will be assessed.
Change From Baseline in estimated Glomerular Filtration Rate (eGFR) | Baseline, Up to Visit 4 (Week 48)
  The change from baseline in eGFR will be assessed by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.
Change From Baseline in Aspartate Transferase (AST) | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Alanine-Amino Transferase (ALT) | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Gamma-Glutamyl Transferase (GGT) | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Alkaline Phosphatase (ALP) | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Total Cholesterol | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Low Density Lypoprotein (LDL) | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in High Density Lypoprotein (HDL) | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Triglycerides | Baseline, Up to Visit 4 (Week 48)
Change From Baseline in Glucose | Baseline, Up to Visit 4 (Week 48)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.